CLINICAL TRIAL: NCT04752475
Title: Lasix for the Prevention of De Novo Postpartum Hypertension: A Randomized Controlled Trial (LAPP Trial)
Brief Title: Lasix for the Prevention of De Novo Postpartum Hypertension
Acronym: LAPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAT2525
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Pregnancy-Induced Hypertension; Postpartum Preeclampsia; Hypertension, Pregnancy-Induced; Hypertension
Keywords: De novo postpartum hypertension; New-onset postpartum hypertension; Lasix; Furosemide
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled clinical trial of 82 women with one or more high-risk factors for de novo postpartum hypertension, randomized to one of two arms: 20 mg PO Lasix (furosemide) daily for 5 days or identical-appearing daily placebo for 5 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Consenting women will be assigned to Lasix (furosemide) or placebo in a 1:1 ratio according to a randomization scheme achieved using a computer generated algorithm. Neither the participant nor the clinical care team will be aware of the allocation arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lasix (furosemide) (Experimental): Furosemide 20 mg, oral, once daily for 5 days
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): Identical-appearing placebo, oral, once daily for 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Furosemide — Furosemide 20 mg pill taken daily for 5 days
  Other Names: Lasix
  Arms: Lasix (furosemide)
Other: Placebo — Identical-appearing placebo pill taken daily for 5 days
  Arms: Placebo

SUMMARY:
Primary objective: To evaluate whether oral furosemide can help prevent de novo postpartum hypertension (new-onset high blood pressure after delivery) by reducing blood pressure after delivery in high-risk women.

Secondary objectives: To evaluate whether oral furosemide administered to high-risk women after delivery can reduce the frequency of postpartum hypertensive episodes, the need for antihypertensive therapy, the risk of postpartum preeclampsia, and the incidence of severe maternal morbidity.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy are one of the leading causes of maternal morbidity and mortality worldwide. The majority of clinical research has focused on pregnancy-related hypertension that develops in the antenatal period, while studies of the incidence, risk factors, and prevention of postpartum hypertension are limited. In particular, there is a paucity of data about the clinical entity known as de novo postpartum hypertension, in which women who are normotensive throughout pregnancy and delivery subsequently go on to develop high blood pressure in the immediate to late postpartum period. Of those with postpartum preeclampsia, 33-69% were normotensive antepartum.

Early identification and treatment of antepartum preeclampsia has been shown to decrease some severe maternal outcomes. Conversely, women with de novo postpartum hypertensive disorders remain among the highest risk for severe maternal morbidity due to decreased surveillance and lack of data regarding preventive therapies and interventions. Evidence from multiple randomized controlled trials have demonstrated a benefit in the use of oral loop-diuretics in decreasing postpartum systolic blood pressure, promoting faster normalization of blood pressure, and decreasing the need for antihypertensive therapy in women with an antenatal diagnosis of preeclampsia. Biological plausibility suggests that loop-diuretic therapy may similarly mitigate the normal physiologic mechanism that has been implicated in the pathogenesis of hypertensive complications after delivery in women at risk for de novo postpartum hypertension.

This study is a double-blind randomized placebo-controlled trial of 82 high-risk women to assess whether treatment with oral Lasix (furosemide) after delivery reduces blood pressure at the time of discharge. Women at high risk for de novo postpartum hypertension will be randomized to a five-day course of either 20 mg oral Lasix (furosemide) or placebo once daily initiated after delivery. Women will be monitored through their routine 2-week and 6-week postpartum visits, during which times hypertensive complications and adverse effects of therapy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women
* No antenatal diagnosis of hypertensive disorder of pregnancy at the time of admission for delivery, defined as existing chronic hypertension diagnosis or documented blood pressure of ≥140 systolic OR ≥90 diastolic on at least 2 occasions at least 4 hours apart prior to delivery admission who do not go on to get magnesium for seizure prophylaxis by the time of delivery
* At least 18 years of age
* English or Spanish speakers
* One or more high risk factors for development of de novo postpartum hypertension

Exclusion Criteria:

* Non-English or Spanish speakers
* Women with a contraindication to diuretic therapy
* Women who have used diuretics in the two weeks prior to delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell S. Miller, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark SL, Belfort MA, Dildy GA, Herbst MA, Meyers JA, Hankins GD. Maternal death in the 21st century: causes, prevention, and relationship to cesarean delivery. Am J Obstet Gynecol. 2008 Jul;199(1):36.e1-5; discussion 91-2. e7-11. doi: 10.1016/j.ajog.2008.03.007. Epub 2008 May 2. PMID 18455140
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Al-Safi Z, Imudia AN, Filetti LC, Hobson DT, Bahado-Singh RO, Awonuga AO. Delayed postpartum preeclampsia and eclampsia: demographics, clinical course, and complications. Obstet Gynecol. 2011 Nov;118(5):1102-1107. doi: 10.1097/AOG.0b013e318231934c. PMID 21979459
- [Background] Filetti LC, Imudia AN, Al-Safi Z, Hobson DT, Awonuga AO, Bahado-Singh RO. New onset delayed postpartum preeclampsia: different disorders? J Matern Fetal Neonatal Med. 2012 Jul;25(7):957-60. doi: 10.3109/14767058.2011.601365. Epub 2011 Aug 16. PMID 21740315
- [Background] Matthys LA, Coppage KH, Lambers DS, Barton JR, Sibai BM. Delayed postpartum preeclampsia: an experience of 151 cases. Am J Obstet Gynecol. 2004 May;190(5):1464-6. doi: 10.1016/j.ajog.2004.02.037. PMID 15167870
- [Background] Sibai BM. Diagnosis, prevention, and management of eclampsia. Obstet Gynecol. 2005 Feb;105(2):402-10. doi: 10.1097/01.AOG.0000152351.13671.99. PMID 15684172
- [Background] Lubarsky SL, Barton JR, Friedman SA, Nasreddine S, Ramadan MK, Sibai BM. Late postpartum eclampsia revisited. Obstet Gynecol. 1994 Apr;83(4):502-5. doi: 10.1097/00006250-199404000-00003. PMID 8134057
- [Background] Bigelow CA, Pereira GA, Warmsley A, Cohen J, Getrajdman C, Moshier E, Paris J, Bianco A, Factor SH, Stone J. Risk factors for new-onset late postpartum preeclampsia in women without a history of preeclampsia. Am J Obstet Gynecol. 2014 Apr;210(4):338.e1-338.e8. doi: 10.1016/j.ajog.2013.11.004. Epub 2013 Nov 7. PMID 24211478
- [Background] Chames MC, Livingston JC, Ivester TS, Barton JR, Sibai BM. Late postpartum eclampsia: a preventable disease? Am J Obstet Gynecol. 2002 Jun;186(6):1174-7. doi: 10.1067/mob.2002.123824. PMID 12066093
- [Background] Ascarelli MH, Johnson V, McCreary H, Cushman J, May WL, Martin JN Jr. Postpartum preeclampsia management with furosemide: a randomized clinical trial. Obstet Gynecol. 2005 Jan;105(1):29-33. doi: 10.1097/01.AOG.0000148270.53433.66. PMID 15625138
- [Background] Veena P, Perivela L, Raghavan SS. Furosemide in postpartum management of severe preeclampsia: A randomized controlled trial. Hypertens Pregnancy. 2017 Feb;36(1):84-89. doi: 10.1080/10641955.2016.1239735. Epub 2016 Nov 11. PMID 27835048
- [Background] Perdigao JL, Lewey J, Hirshberg A, et al. LB 4: Furosemide for Accelerated Recovery of Blood Pressure Postpartum: a randomized placebo controlled trial (FoR BP). American Journal of Obstetrics & Gynecology. 2020;222(1):S759-S760.
- [Background] Atterbury JL, Groome LJ, Hoff C. Blood pressure changes in normotensive women readmitted in the postpartum period with severe preeclampsia/eclampsia. J Matern Fetal Med. 1996 Jul-Aug;5(4):201-5. doi: 10.1002/(SICI)1520-6661(199607/08)5:43.0.CO;2-O. PMID 8796794
- [Background] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lasix (Furosemide) | Placebo
Started | 41 | 41
Completed | 40 | 40
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data collected and analyzed for 80 of the 82 participants - 2 participants who initially consented to participate in the trial subsequently withdrew prior to discharge from delivery hospitalization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lasix (Furosemide) | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Customized [Count of Participants; unit: Participants]
  age < 35 | 17 | 12 | 29
  age >= 35 | 23 | 28 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 22 | 27 | 49
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 9 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 9 | 9
  Black or African American | 10 | 0 | 10
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 10 | 25
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure (MAP)
Description: Difference in MAP averaged over the 24 hours prior to discharge or the 24 hours prior to antihypertensive therapy initiation (whichever occurs first)
Time Frame: 24 hours prior to discharge through discharge, up to 7 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 40
mmHg | 88.9 (7.4) | 86.8 (7.1)

2. Secondary Outcome: Time to Discharge
Description: Time until discharge from the hospital
Time Frame: Randomization through discharge, up to 7 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 40
days | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]

3. Secondary Outcome: Rate of de Novo Postpartum Preeclampsia
Description: Number of participants who develop de novo postpartum hypertension. This outcome was assessed at Discharge (up to 7 days), 2 weeks postpartum, and 6 weeks postpartum. Data is reported at 6 weeks postpartum.
Time Frame: Discharge (up to 7 days), 2 weeks postpartum, 6 weeks postpartum
Population: 1 participant in the Placebo Arm (who completed Primary Outcome) withdrew from the study before the Secondary Outcome data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 5 | 3

4. Secondary Outcome: Percent of Recorded Blood Pressures That Are Elevated
Description: Percent of recorded blood pressures that are elevated (>140 systolic OR >90 diastolic).
Time Frame: Discharge (up to 7 days), 2 weeks postpartum, 6 weeks postpartum
Population: 1 participant in the Placebo Arm withdrew from the study before the Secondary Outcome data was collected.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
percent
  Discharge | 4 [0 to 9] | 0 [0 to 6]
  2 weeks postpartum | 8 [5 to 17] | 5 [2 to 13]
  6 weeks postpartum | 8 [4 to 17] | 5 [2 to 9]

5. Secondary Outcome: Rate of Magnesium Sulfate Administration
Description: Number of participants who receive intravenous magnesium sulfate for seizure prophylaxis. This outcome was assessed at Discharge (up to 7 days), 2 weeks postpartum, and 6 weeks postpartum. Data is reported at 6 weeks postpartum.
Time Frame: Discharge (up to 7 days), 2 weeks postpartum, 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 2 | 2

6. Secondary Outcome: Rate of Initiation of Antihypertensives
Description: Number of participants receiving intravenous antihypertensive therapy and initiated on oral hypertensive therapy. This outcome was assessed at Discharge (up to 7 days), 2 weeks postpartum, and 6 weeks postpartum. Data is reported at 6 weeks postpartum.
Time Frame: Discharge (up to 7 days), 2 weeks postpartum, 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 4 | 3

7. Secondary Outcome: Rate of Severe Maternal Morbidity
Description: Number of participants experiencing severe maternal morbidity (e.g. seizure, stroke, Posterior reversible encephalopathy syndrome (PRES), death, etc.) This outcome was assessed at Discharge (up to 7 days), 2 weeks postpartum, and 6 weeks postpartum. Data is reported at 6 weeks postpartum.
Time Frame: Discharge (up to 7 days), 2 weeks postpartum, 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 0 | 1

8. Secondary Outcome: Rate of Triage or Emergency Department (ED) Presentation/Readmission
Description: Number of participants who experienced triage or ED presentation/readmission for hypertensive-related complaints. This outcome was assessed at 2 weeks postpartum and 6 weeks postpartum. Data is reported at 6 weeks postpartum.
Time Frame: 2 weeks postpartum, 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants | 4 | 2

9. Secondary Outcome: Breastfeeding Continuation Rate
Description: Number of participants continuing to breastfeed of those who initiated breastfeeding after delivery. This outcome was assessed at Discharge (up to 7 days), 2 weeks postpartum, and 6 weeks postpartum. Data is reported at 2 weeks and 6 weeks postpartum.
Time Frame: 2 weeks postpartum, 6 weeks postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lasix (Furosemide) | Placebo
Number analyzed (Participants) | 40 | 39
Participants
  2 weeks | 5 | 5
  6 weeks | 7 | 5

ADVERSE EVENTS:
Time Frame: Up to 6 weeks postpartum
Arm/Group | Lasix (Furosemide) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04752475/Prot_SAP_000.pdf